CLINICAL TRIAL: NCT05071781
Title: The Effect of Corticotropin Release Hormone on Duodenal Markers and Gastric Sensorimotor Function in Healthy Volunteers
Brief Title: Effect of CRH on Duodenal Markers and Gastric Sensorimotor Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S65020
Record Dates: First submitted 2021-08-16; First posted 2021-10-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: GI Motility Disorder
Keywords: cortisol releasing hormone; 3.1 Functional dyspepsia

STUDY DESIGN:
Intervention Model Description: To assess the effect of the CRH on on duodenal mast cell count, eosinophil count, immune activation and mucosal permeability, gastric accommodation, gastric sensitivity to distension and gastric emptying time, an interventional study will be conducted in 20 healthy subjects. The study is designed as a double-blind randomized crossover study with at least 7 days between the different study days.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cortisol releasing hormone group (Active Comparator): HVs will start with CRH infusion.
  Interventions: Drug: Corticotropin-release hormone
- Placebo (sodium choride) group (Placebo Comparator): HVs will start with NaCl 0.9% (placebo) infusion
  Interventions: Drug: Corticotropin-release hormone

INTERVENTIONS:
Drug: Corticotropin-release hormone — intravenous CRH (100 µg)
Drug: Corticotropin-release hormone — a bolus dose (CRH 100 µg or placebo) will be administered, followed by a continuous infusion (CRH 1 µg/kg/h or placebo)

SUMMARY:
In the present study, during Part 1, after a baseline gastroduodenoscopy, the investigators will perform a gastroduodenoscopy twice, to take duodenal biopsies before and 2 hours after administration of CRH/placebo. The investigators will measure mucosal integrity and markers of immune activation as outlined in Parts A and B, and will use transmission electron microscopy to evaluate mast cell and eosinophil degranulation. After an interval period of at least 1 week, CRH or placebo will be administrated again in a crossover fashion.

As a complementary study, the investigators will also test the effect of ex vivo mast cell blockade by lodoxamide to evaluate whether mast cells are involved in the hypothesized effect of CRH on duodenal permeability.

In a second part of this study, Part 2, the investigators will perform a gastric barostat, to measure the gastric accommodation and sensitivity to distension, and a carbon-13-octanoic acid breath test to measure the gastric emptying time after administration of CRH/placebo.

Healthy volunteers will have the option to choose to which part of the study (part 1 or 2) they wish to participate. They can also choose to cooperate to both study parts if preferred.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant has been obtained prior to any screening procedures
2. Women of child-bearing potential agree to apply a highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
3. Healthy volunteers
4. Subjects aged 18-55 years old (55y included).
5. Male or female subjects.
6. Subjects who are capable to understand the study and the questionnaires, and to comply with the study requirements.

Exclusion Criteria:

1. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
2. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
3. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
4. Presence of a history of gastrointestinal surgery other than appendectomy
5. Presence of organic or functional gastrointestinal disease
6. Presence of gastro-intestinal symptoms
7. Major psychiatric disorder such as major depression
8. Presence of any disease affecting the gastrointestinal tract or hepatobiliary system.
9. History of allergic reaction to CRH
10. BMI equal to 30 mg/kg² or higher.
11. Use of drugs included in this list:

    1. Opioids (unless short intake for acute pain and > 1month ago)
    2. Amitriptyline or mirtazapine; other antidepressants are allowed if the HV is on a stable dose and the drug is not combined with other antidepressants.
    3. Corticosteroids
    4. Antihistaminic drugs (last 2 weeks)
    5. Proton pump inhibitors (last 2 weeks)
    6. Disodiumchromoglycate or other mast cell stabilizers (last 2 weeks)
    7. Leukotriene receptor antagonists (last 2 weeks)
    8. NSAIDs (last 2 weeks)
    9. Antibiotics (last 2 months)
    10. Probiotics (last 2 weeks)
    11. Other medication: to be discussed with physician

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
The effect of corticotrophin release hormone (CRH) on duodenal mast cell count | 2 hours after CRH/placebo
  Duodenal mast cells (c-kit) will be counted per mm2 via stained duodenal biopsy sections.
The effect of CRH on sensitivity to gastric distention (part 2) | 30 minutes after CRH/placebo
  Visceral sensitivity will be measured by barostat. Discomfort threshold will be defined as the first level of pressure and the corresponding volume that provokes discomfort. Pressure thresholds will be expressed both as pressures relative to minimal distending pressure and as absolute pressures.

SECONDARY OUTCOMES:
The effect of CRH on duodenal eosinophilia | 2 hours after CRH/placebo
  Duodenal eosinophils (H&E) will be counted per mm2 via stained duodenal biopsy sections.
The effect of CRH on duodenal mucosal permeability | 2 hours after CRH/placebo
  Duodenal mucosa permeability on duodenal biopsies using adapted mini-Ussing chambers
The effect of CRH on gastric emptying time | 30 minutes after CRH/placebo
  Gastric emptying time in minutes t (1/2) will be measured by 13C-octanoic acid breath test.
The effect of CRH on gastric accommodation | 30 minutes after CRH/placebo
  Gastric accommodation will be measured by barostat. Accommodation to a meal will be expressed as the average increase in intragastric volume during the first 4 postprandial hours.
The effect of CRH on gastroduodenal symptoms. | Every 15 minutes during CRH/placebo infusion for 4 hours
  Assessments using Visual Analog Score for GI symptoms which including pain, nausea, bloating, vomiting.
The effect of CRH on salivary cortisol level | Right before CRH/placebo injection, 15, 30, 60, 120 minutes after injection
  Salivary cortisol level in nmol/L during placebo or CRH infusion

CONTACTS AND LOCATIONS:
Locations (1):
- I-Hsuan Huang, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
The Trial will be conducted in compliance with the requirements of the EU General Data Protection Regulation 2016/679 (GDPR), the relevant Belgian laws implementing the GDPR including the Belgian Privacy Act of 30 July 2018 on the protection of privacy in relation to the processing of personal data. Any collection, processing and disclosure of personal data, such as participant health and medical information is subject to compliance with the aforementioned personal data protection laws.